CLINICAL TRIAL: NCT01679535
Title: A Nutrition/Hygiene Education Program for the Prevention of Child Malnutrition in Rural Kenya
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Not an applicable clinical trial (ACT).
Sponsor: University of New Mexico (Other)
Collaborators: University of Nairobi (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: TOMEDI-12-049
Record Dates: First submitted 2012-08-29; First posted 2012-09-06 (Estimated); Last update posted 2024-03-12 (Actual); Status verified 2024-03

CONDITIONS: Child Nutrition Disorders
Keywords: Infant nutrition disorder; Child nutrition disorders; Malnutrition; Protein-energy malnutrition
MeSH Terms: conditions — Child Nutrition Disorders; Infant Nutrition Disorders; Malnutrition; Protein-Energy Malnutrition | interventions — Nutritional Status

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intervention (Experimental): nutrition and hygiene education by community health workers
  Interventions: Behavioral: nutrition and hygiene education

INTERVENTIONS:
Behavioral: nutrition and hygiene education — Monthly education sessions about child feeding and hygiene for mothers of young children, conducted by local Kenyan community health workers

SUMMARY:
This study will determine if an education program about hygiene and child feeding practices, taught by local village community health workers, will improve child growth and decrease the prevalence of childhood malnutrition in a rural region of Kenya.

ELIGIBILITY:
Inclusion Criteria:

* Child of a mother living in the catchment area of the study who delivered during the enrollment period

Ages: 1 Month to 6 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 246 (Actual)
Dates: Start 2011-11 (Actual); Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
malnutrition prevalence | Measured when children are 24 months of age
  Child malnutrition rates, as measured by the prevalence of underweight, wasting, and growth stunting of the children in each group

SECONDARY OUTCOMES:
Child growth | Measured when children are 24 months of age
  Child growth as measured by change in z score of the children in each group

OTHER OUTCOMES:
Prevalence of diarrhea | Prevalence assessed when children reach 24 months of age

CONTACTS AND LOCATIONS:
Overall Officials: Angelo J Tomedi, MD, Principal Investigator — University of New Mexico
Locations (1):
- University of New Mexico, Albuquerque, New Mexico, United States

REFERENCES:
- [Result] Black RE, Allen LH, Bhutta ZA, Caulfield LE, de Onis M, Ezzati M, Mathers C, Rivera J; Maternal and Child Undernutrition Study Group. Maternal and child undernutrition: global and regional exposures and health consequences. Lancet. 2008 Jan 19;371(9608):243-60. doi: 10.1016/S0140-6736(07)61690-0. No abstract available. PMID 18207566
- [Result] Bhutta ZA, Ahmed T, Black RE, Cousens S, Dewey K, Giugliani E, Haider BA, Kirkwood B, Morris SS, Sachdev HP, Shekar M; Maternal and Child Undernutrition Study Group. What works? Interventions for maternal and child undernutrition and survival. Lancet. 2008 Feb 2;371(9610):417-40. doi: 10.1016/S0140-6736(07)61693-6. PMID 18206226
- [Result] Dewey KG, Adu-Afarwuah S. Systematic review of the efficacy and effectiveness of complementary feeding interventions in developing countries. Matern Child Nutr. 2008 Apr;4 Suppl 1(Suppl 1):24-85. doi: 10.1111/j.1740-8709.2007.00124.x. PMID 18289157